CLINICAL TRIAL: NCT06393959
Title: Comparison of Pulsed Radiofrequency Stimulation Versus Dexamethasone Applied to the Caudal Epidural Space for the Relief of Lumbar Spinal Stenosis Symptoms
Brief Title: Relief of Lumbar Spinal Stenosis Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Supervisor Investigator, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Spinal Stenosis
Record Dates: First submitted 2024-04-27; First posted 2024-05-01 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Spinal Stenosis Lumbar; Low Back Pain
Keywords: Pulsed Radiofrequency Treatment; Lomber spinal Stenosis; Caudal epidural steroid injection
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pulsed radiofrequency group (Active Comparator): Caudal epidural pulsed radiofrequency for lumbar spinal stenosis
  Interventions: Procedure: Caudal epidural pulsed radiofrequency
- steroid enjection grroup (Active Comparator): Caudal epidural steroid enjection for lumbar spinal stenosis
  Interventions: Procedure: Caudal epidural steroid enjection

INTERVENTIONS:
Procedure: Caudal epidural pulsed radiofrequency — The patient lied in prone position. After cutaneous and subcutaneous anesthesia with 3 ml of 2% lidocaine, a 22- gauge 150-mm RF cannula with 20 mm active tip was advanced through the sacrococcygeal ligament into the caudal epidural space under floroscopic guidence. A few milliliters contrast was injected to observe the expansion of the epidural space. After correct needle placement was confirmed, an electrode was connected to the cannula, and stimulation was conducted with impedance measured between 250 and 350 Ohms A different sensation or feeling such as fullness, impression, tingling, pulling or plethora at the rectal and/or coccygeal region was observed by the patients when 50 Hz was applied with 0,4 to 0,7 V sensory stimulation. No leg muscle contraction was observed with 2 Hz motor stimulation at 2 V. PRF was performed for 600 s at 5 Hz using a 5-ms pulse width at 55 V, avoiding electrode tip temperatures above 42 C.
  Arms: pulsed radiofrequency group
Procedure: Caudal epidural steroid enjection — The patient lied in prone position and aseptic techniques were adopted. After cutaneous and subcutaneous anesthesia with 3 ml of 2% lidocaine, a spinal needle was advanced through the sacrococcygeal ligament into the caudal epidural space under fluoroscopic guidance. The needle tip was confirmed by negative aspiration for blood or cerebrospinal fluid, then a few milliliters of contrast was injected to observe the expansion of the epidural space. After correct needle placement was confirmed, a total of 10 ml mixture of saline and 8 mg dexametzone was administered into the epidural space.
  Arms: steroid enjection grroup

SUMMARY:
The aim of this study was to compare the efficacy of caudal epidural steroid injection and caudal epidural pulsed radiofrequency stimulation in the relief of symptoms of lumbar spinal stenosis.

This evaluation used the numerical rating scale (NRS) to assess pain relief and the Medication Quantification Scale III (MQS III) to assess the effectiveness of the interventions on medication consumption. The rates of adverse events related to the interventions were also compared.

DETAILED DESCRIPTION:
Low back pain (LBP) is one of the leading causes of disability worldwide. Lumbar spinal stenosis is one of the three most common diagnoses of lower back and leg pain, along with intervertebral disc herniation and degenerative spondylolisthesis. Numerous treatment modalities have been proposed for the management of lumbar spinal stenosis, including drug therapy and complex surgical fusion. Epidural injections are a nonsurgical intervention commonly used in the treatment of spinal stenosis. Saline, local anesthetics, steroids, hylaze, platelet-rich plasma, and pulsed radiofrequency (PRF) administered to the caudal epidural space have been reported to be effective in the treatment of pain.

Among these, caudal epidural PRF has been applied in a limited number of chronic painful conditions (failed back surgery syndrome, chronic distal symmetrical polyneuropathy, postherpetic neuralgia, and coccygodynia), and no randomized controlled studies have been conducted. PRF produces a nonthermal effect that modulates the transmission of pain signals by delivering a short-term high-voltage electric current to the target nerve. RFT provides a continuous current that heats the target tissue and causes coagulation necrosis in nerves.

The primary aim of this study was to compare the efficacy of caudal epidural RFT and caudal epidural steroid injections in patients with lumbar spinal stenosis. The secondary aim was to determine the effects of the interventions on drug consumption and interventional safety, based on adverse events.

A total of at least 50 patients will be enrolled for comparison, with 25 in each group. NRS and MQS III scores will be compared both within and between groups before and 1, 2, and 3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

Among the patients with lumbar spinal stenosis findings and narrowing of the spinal canal detected by examination and imaging methods, those whose back and leg pain persists for at least 3 months

Exclusion Criteria:

Previous lumbar surgery, pregnancy, history of ongoing malignant disease, autoimmune diseases, active infection of the injection site, hematologic disorders, antiplatelet drug use

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-07-19 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
Numerical rating scale (NRS) | Change from baseline to 1st,2nd and 3th month after treatment
  NRS is a scale that can be used measuring pain. Scores range from 0 (no pain) to 10 (the worst pain)

SECONDARY OUTCOMES:
The Medication Quantification Scale III (MQS III) | Change from baseline to 1st,2nd and 3th month after treatment
  The MQS III is a validated tool in medical research that quantifies medication regimens by assigning a numerical value to each medication based on its class, dosage, and associated risks. This scale aids clinicians and researchers in tracking changes in pain levels throughout a treatment course or study, providing an objective measure of medication consumption and its potential negative impact.

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Taylan T Akkaya, Prof, Principal Investigator — Department of Algology, Ankara Etlik City Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Damla Yürük, Ankara, Türkiye
  - Ankara Etlik City Hospital, Ankara, Yenimahalle